CLINICAL TRIAL: NCT02830685
Title: Prospective Multicentric Randomized Comparison of an Acellular Dermal Matrix Versus a Synthetic Mesh in DIRECT-TO-IMPLANT (DTI) Pre-pectoral Implant Based Breast Reconstruction
Brief Title: Pre-pectoral Breast Reconstruction PART 1
Acronym: PreBRec
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Kovacs, MD, PhD, Guy's and St Thomas' NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCTBU012016
Record Dates: First submitted 2016-06-28; First posted 2016-07-13 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
Keywords: pre-pectoral breast reconstruction; subcutaneous breast reconstruction
MeSH Terms: conditions — Breast Neoplasms | interventions — Diffusion Tensor Imaging

ARMS (2):
- Direct-To-Implant A (Active Comparator): DTI with Acellular Dermal Matrix (CELLIS® Breast), pre-pectoral, subcutaneous direct-to-implant breast reconstruction with the aid of an Acelluar Dermal Matrix (ADM)
  Interventions: Device: DTI with Acellular Dermal Matrix (CELLIS® Breast)
- Direct-To-Implant B (Experimental): DTI with Titanium Coated Polypropylene Mesh (TiLOOOP® Bra), pre-pectoral, subcutaneous direct-to-implant breast reconstruction with the aid of a titanium coated polypropylene mesh
  Interventions: Device: DTI with Titanium Coated Polypropylene Mesh (TiLOOOP® Bra)

INTERVENTIONS:
Device: DTI with Acellular Dermal Matrix (CELLIS® Breast) — After conservative mastectomy, a pre-pectoral subcutaneous reconstruction with definitive implant will be performed using an ADM (CELLIS® Breast), either completely covering the implant or simply covering the anterior surface of it. The implant could be of any shape, material and texture available with no restriction. After at least 6 months, a fat grafting procedure, using a wash and filter principle for fat handling, will be performed over the implant.
  Other Names: Pre-pectoral Direct-to-implant with ADM, fat grafting
  Arms: Direct-To-Implant A
Device: DTI with Titanium Coated Polypropylene Mesh (TiLOOOP® Bra) — After conservative mastectomy, a pre-pectoral subcutaneous reconstruction with definitive implant will be performed using a TCPM (TiLOOOP® Bra), either completely covering the implant or simply covering the anterior surface of it.The implant could be of any shape, material and texture available with no restriction. After at least 6 months, a fat grafting procedure, using a wash and filter principle for fat handling, will be performed over the implant.
  Other Names: Pre-pectoral Direct-to-implant with TCPM, fat grafting
  Arms: Direct-To-Implant B

SUMMARY:
The rationale for present trial conception and design moves forward from the assumption that a subcutaneous, pre-pectoral reconstruction by means of soft tissue replacement devices is feasible, safe and giving rewarding results when compared to the standard retro-pectoral technique. Ahead of that, the trial aims to test if there is a difference in the outcomes between a biological and a synthetic material when placed as a support under the mastectomy skin flaps, both in terms of immediate complications and of long-term results.

DETAILED DESCRIPTION:
This phase III randomized clinical trial will compare direct-to-implant pre-pectoral breast reconstruction with different supportive materials:

the trial will comprise two arms: A-PRE-PECTORAL technique with a biological Acellular Dermal Matrix (ADM) prosthesis coverage and support + FAT GRAFTING VS B-PRE-PECTORAL technique with a synthetic Titanium Coated Polypropylene Mesh (TCPM) prosthesis coverage and support + FAT GRAFTING

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria will entail cases of conservative mastectomies (skin-sparing mastectomy SSM

* Nipple-sparing mastectomy NSM and skin-reducing mastectomy SRM)
* Prophylactic and therapeutic.

Included patients baseline characteristics will be:

* Age 18-80 years old
* BMI between 18.5 and 35.
* Former smokers (up until 3 weeks before surgery)
* Hypertension at oral medications
* Diabetes
* Previous breast surgery
* Previous breast and chest wall radiation therapy will be allowed.

Exclusion Criteria:

* T4 and metastatic breast cancers
* Obese patients (BMI over 35)
* Currently smoking patients (within 3 weeks before surgery)
* Refusal to sign the consent
* Severe comorbidities requiring a chronic therapy (renal failure, heart failure, cardiovascular diseases, pulmonary diseases, hepatic diseases, and metabolic diseases).

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-07 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Rate in percentage of surgical complications | up to 6 months
  Surgical outcomes within the first six months from mastectomy and IBBR will be evaluated with the statistical difference in percentage rate of complicated and non complicated patients between the two groups. Complications will be the following:
  surgical site infection (any infection requiring an antibiotic therapy, either oral or intravenous), wound dehiscence, seroma (any fluid collection requiring aspiration for more than a month from mastectomy), nipple/skin necrosis (either partial or complete), hematoma, red breast syndrome, with their reintervention rate, all in percentages.
Rate in percentage of technique failure | up to 6 months
  The failure rate will be assessed considering the statistical difference in percentage rate of removed implants among total number and comparing them between the two arms: in other words the prostheses (implants) loss rate (reinterventions with prosthesis removal).

SECONDARY OUTCOMES:
Objective quality of life assessment with Baker scale for capsular contracture | at 2 years from mastectomy
  Quality of life outcomes at 2 years from mastectomy and at least 3 months after completion of the reconstructive step included in the protocol (one fat grafting procedure) will entail first of all an objective evaluation: such evaluation will be performed with the the scoring of capsular contracture rate, including assessment of the reintervention rate for amelioration or for a reconstructive strategy change, comparing the two arms.
Objective quality of life assessment with cosmetic evaluation on pictures with a Likert scale scoring | at 2 years from mastectomy
  In addition another objective analysis will include a third party objective evaluation, carried out by a group of a surgeon, a nurse and a lay person from a different center from that one where every single case was performed. This third party evaluation will assess the cosmetic outcome based on medical photographic files. Scores from this ranking will be compared between the two groups.
Subjective quality of life assessment using the BREAST-Q questionnaire (Memorial Sloan-Kettering Cancer Center and The University of British Columbia © 2006, all rights reserved). | at 2 years from mastectomy
  Quality of life outcomes at 2 years from mastectomy and at least 3 months after completion of the reconstructive step included in the protocol (one fat grafting procedure) will entail also a subjective evaluation: such evaluation will be carried out using the BREAST-Q questionnaire. Scores will be transformed in a 100 scale and compared as median between the two groups.

OTHER OUTCOMES:
Cost-efficiency analysis with comparison of costs in money of the two different procedures and following possible adjunctive costs for reintervention in case of complications | at 3 years from mastectomy
  A long-term evaluation of costs will be carried out for all cases, considering procedures, hospitalizations, days off from work and long-term readmission and revision surgeries. These data will be compared between arms and with every other type of reconstruction. A specific similar analysis will be conducted on irradiated cases comparing with non irradiated.
Rate in percentage of surgical complications in the sub-group of irradiated patients | at 3 years from mastectomy
  An analysis of the subgroup of patients with a previous breast irradiation or a post-mastectomy radiation therapy will be carried out considering short-term complications leading to failures and long-term complications leading to change in reconstruction strategy.

CONTACTS AND LOCATIONS:
Locations (1):
- Breast Unit Surgery, Guy's and St Thomas' Hospital NHS Trust, London, United Kingdom